CLINICAL TRIAL: NCT04790552
Title: The Effects of Fast Bar on Facilitating Prolonged Fasting - a Randomized, Controlled, Parallel-arm Study
Brief Title: Effects of Fast Bar on Intermittent Fasting
Acronym: FastBar2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L-Nutra Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LN002; 20210458 (Other: WIRB)
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Fasting
Keywords: Fast Bar; Intermittent fasting; Ketone bodies; ß-hydroxybutyrate
MeSH Terms: conditions — Fasting; Intermittent Fasting | interventions — Meals; Angptl4 protein, mouse; Receptors, Catecholamine; Coffee; Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fast Group (Active Comparator): Subjects will be asked to consume a standardized ready-to-eat dinner meal before 5 pm on day 1. Subjects will fast overnight for approximately 19 hours.
  Interventions: Other: Dinner; Other: Fasting
- Night Bar Group (Experimental): Subjects will be asked to consume a standardized ready-to-eat dinner meal before 5 pm on day 1. Subjects will consume a Fast Bar 3 hours after the dinner and then fast overnight. Subjects will fast overnight for approximately 15 hours and then consume a Fast Bar with coffee on day 2.
  Interventions: Other: Dinner; Other: Fasting; Other: Fast Bar
- Bar + Coffee Group (Experimental): Subjects will be asked to consume a standardized ready-to-eat dinner meal before 5 pm on day 1. Subjects will fast overnight for approximately 15 hours and then consume a Fast Bar with coffee on day 2.
  Interventions: Other: Dinner; Other: Fasting; Other: Bar with Coffee
- Bar + Tea Group (Experimental): Subjects will be asked to consume a standardized ready-to-eat dinner meal before 5 pm on day 1. Subjects will fast overnight for approximately 15 hours and then consume a Fast Bar with tea on day 2.
  Interventions: Other: Dinner; Other: Fasting; Other: Bar with Tea

INTERVENTIONS:
Other: Dinner — Study subjects will consume a standardized ready-to-eat meal as dinner.
Other: Fasting — Subjects will be asked to fast overnight for approximately 15 hours.
Other: Fast Bar — Subjects will be asked to consume a Fast Bar.
  Arms: Night Bar Group
Other: Bar with Coffee — Subjects will be asked to consume a Fast Bar with coffee.
  Arms: Bar + Coffee Group
Other: Bar with Tea — Subjects will be asked to consume a Fast Bar with tea.
  Arms: Bar + Tea Group

SUMMARY:
This study evaluates how Fast Bar(TM), a specially formulated energy bar, when consumed with coffee or tea, affects the physiological condition in participants after an overnight fasting. Participants will fast for 19 hours (Fast Group), consume a Fast Bar in the night (Night Bar Group) or in the morning (Bar+Coffee and Bar+Tea Groups) after an approximately 15-hour overnight fasting. Participants will be assessed for physiological parameters associated with fasting.

DETAILED DESCRIPTION:
Interest in fasting-based programs (i.e. intermittent fasting) for improvement of health and longevity continues to grow. The short-term fasting (e.g. 12 to 48 hours in duration) utilized in many intermittent fasting programs are considered safe, but some individuals may find them subjectively difficult. As such, the question of whether the benefits of fasting can be obtained while small amounts of food are consumed is of substantial interest.

One commercially available product that is designed to be consumed during periods of intermittent fasting is the Fast Bar™, which stems out of the well-researched fasting-mimicking diet to assist prolonged fasting. The unique formulation of the Fast Bar™ is hypothesized to minimize deviations in metabolic biomarkers associated with a fasting state. This may ease the burdens associated with extended period of fasting. The objective of this study is to evaluate the metabolic and subjective effects of Fast Bar, when consumed with coffee or tea, after a prolonged period of fasting.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent;
* Ability and willingness to use Zoom teleconference;
* Ability and willingness to perform the study tests and adhere to study protocol to the best of the participant's knowledge;
* 18-65 years of age (inclusive) at screening;
* BMI 20-35 kg/m2 (inclusive) at screening;
* In good health (as determined by medical history to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days);
* Habitual breakfast eater (determined with a screening survey: number of breakfasts per week ≥4.

Exclusion Criteria:

* Has any medical disease or condition that, in the opinion of the principal investigator (PI) or appropriate study personnel, precludes study participation* (*Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial);
* History of gastric bypass (based on medical history provided at screening);
* Under medications aimed at keeping blood glucose under control (based on medical history provided at screening);
* Type 1 diabetes (based on medical history provided at screening);
* Taking insulin, insulin analogs, or octreotide (based on medical history provided at screening);
* Food allergies which would make the subject unable to consume the food provided (based on medical history and information provided at screening) (participants will be asked to review the ingredient lists for the dinner meal and the Fast BarTM, and to state that they are not allergic to the ingredients to the best of their knowledge);
* Women who are pregnant;
* Alcohol dependency (alcohol intake greater than two drinks per day for women and three drinks per day for men) (based on medical history and information provided at screening).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Ketone level | 3 hours after consuming the study foods (Fast Bar with coffee or tea)
  Blood ketone (ß-hydroxybutyrate, BHB) level (mg/dL) will be measured with a Abbott Precision Xtra Blood Glucose and Ketone Monitoring Kit.
Ketone Area Under the Curve | BHB Area Under the Curve between 0 to 4 hours after consuming the study foods
  Blood ketone (ß-hydroxybutyrate, BHB) area under the curve (AUC) will be measured with a Abbott Precision Xtra Blood Glucose and Ketone Monitoring Kit on 0, 1, 2, 3, and 4 hours after consuming the study foods.
Glucose Area Under the Curve | Glucose Area Under the Curve between 0 to 4 hours after consuming the study foods
  Blood glucose area under the curve (AUC) will be measured with a Abbott Precision Xtra Blood Glucose and Ketone Monitoring Kit on 0, 1, 2, 3, and 4 hours after consuming the study foods

SECONDARY OUTCOMES:
Food evaluation | 1 hour after consuming the study foods
  Food Evaluation Questionnaire will be used to assess the subjective evaluation of the study foods. Evaluation will be performed on a Likert Scale from 1 to 7.
Self-evaluation | 1 hour after consuming the study foods
  Self-evaluation Questionnaire will be used to assess the huger and other side-effects associated with a 15-hour overnight fasting. Evaluation will be performed on a Likert Scale from 1 to 7.

CONTACTS AND LOCATIONS:
Overall Officials: William Hsu, MD, Principal Investigator — L-Nutra Inc
Locations (1):
- L-Nutra Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No